CLINICAL TRIAL: NCT02432326
Title: A Phase Ib Clinical Study of BBI608 and BBI503 Administered in Combination to Adult Patients With Advanced Solid Tumors
Brief Title: A Study of BBI608 and BBI503 Administered in Combination to Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBI401-101
Record Dates: First submitted 2015-04-28; First posted 2015-05-04 (Estimated); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Cancer; Advanced Solid Tumors
Keywords: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — napabucasin

ARMS (1):
- Arm A (Experimental)
  Interventions: Drug: BBI608; Drug: BBI503

INTERVENTIONS:
Drug: BBI608 — The BBI608 starting dose is 240 mg twice daily (480 mg total daily). Dose will be decreased to 160 mg twice daily (320 mg total daily) at modification level 2 and 80 mg twice daily (160 mg total daily) at modification level 3. For BBI608 once daily dosing, doses at starting level and modification level 1 are 240 mg once daily, and 480 mg once daily at escalated levels. Dose will be decreased to 160 mg once daily at modification level 2 and 80 mg once daily at modification level 3.
  Other Names: Napabucasin; BB608; BBI-608
Drug: BBI503 — The BBI503 starting dose is 200 mg once daily. Dose at modification level 1 to 3 will be 100 mg once daily.
  Other Names: BB503; BBI-503

SUMMARY:
This is an open label, multi-center, phase 1 study of BBI608 and BBI503 administered orally in combination to patients with advanced solid tumors. The primary goal is to determine the safety, tolerability, and recommended phase II dose (RP2D) of the combination regimen.

ELIGIBILITY:
Inclusion Criteria

1. Signed written informed consent must be obtained and documented according to International Conference on Harmonisation (ICH) and local regulatory requirements
2. A histologically or cytologically confirmed solid tumor that is metastatic, unresectable, or recurrent and for which standard therapies do not exist or are no longer effective

   a. Patients must not be considered eligible for a potentially curative resection
3. ≥ 18 years of age
4. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Male or female patients of child-producing potential must agree to use contraception or avoidance of pregnancy measures during the study and for 30 days after the last dose
7. Females of childbearing potential must have a negative serum pregnancy test
8. Aspartate transaminase (AST) < 2.5 x upper limit of normal (ULN) and alanine transaminase (ALT) ≤ 2.5 × ULN.

   1. Patients who do not have hepatocellular carcinoma but who have liver lesions or liver metastases may be eligible if they have AST < 3.5 x ULN and AST < 3.5 x ULN if agreed upon by the investigator and medical monitor for the sponsor.
   2. Patients with hepatocellular carcinoma may be eligible provided they have AST and ALT that are ≤ 5.0 x ULN.
9. Hemoglobin (Hgb) ≥ 9 g/dL
10. Total bilirubin ≤ 1.5 × ULN. Patients with liver lesions who do not have hepatocellular carcinoma and who have a total bilirubin ≤ 2.0 x ULN may be eligible if agreed upon by the investigator and medical monitor for the sponsor.

    1. Patients with hepatocellular carcinoma may be eligible provided they have total bilirubin ≤ 3.0 x ULN and are considered Child-Pugh Class A or Child-Pugh Class B7 (Child-Pugh Class B with a total Child-Pugh score not to exceed 7).
    2. Patients with Gilbert's syndrome uncomplicated by other liver disease may be eligible if agreed upon by the investigator and medical monitor for the sponsor.
11. Creatinine ≤ 1.5 × ULN or, for patients with creatinine levels above institutional upper limit of normal, creatinine clearance must be > 60 mL/min/1.73 m^2.
12. Absolute neutrophil count ≥ 1.5 x 10^9/L
13. Platelets ≥ 100 x 10^9/L; patients with hepatocellular carcinoma may enroll provided they have a platelet count ≥ 75 x 10^9/L.
14. Life expectancy ≥ 3 months

Exclusion Criteria

1. Anti-cancer chemotherapy, radiotherapy, immunotherapy, or investigational agents within 7 days of first dose of BBI608 and BBI503. Patients may begin BBI608 and BBI503 on a date determined by the investigator and medical monitor for the sponsor after a minimum of 7 days since last receiving anti-cancer treatment, provided that all treatment-related adverse effects have resolved or have been deemed irreversible
2. Surgery within 4 weeks prior to first dose
3. Any known untreated brain metastases. Treated subjects must be stable 4 weeks after completion of treatment for brain metastases and image documented stability is required. Patients must have no clinical symptoms from brain metastases and must be either off of steroids or on a stable dose of steroids for at least 2 weeks prior to protocol enrollment. Patients with known leptomeningeal metastases are excluded, even if treated
4. Pregnant or breastfeeding
5. Significant gastrointestinal disorder(s) (e.g., active Crohn's disease or ulcerative colitis, or a history of extensive gastric resection and/or small intestinal resection) such that absorption of oral medications is impaired.
6. Unable or unwilling to swallow BBI608 and/or BBI503 capsules daily
7. Prior treatment with either BBI608 or BBI503
8. Uncontrolled concurrent illness including, but not limited to ongoing or active infection, clinically significant non-healing or healing wounds, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or on mild exertion), uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements
9. Subjects with a history of another primary cancer, with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; and c) other primary solid tumors (with no known active disease present) that, in the opinion of the investigator, will not affect patient outcome in the setting of the current diagnosis

   1. Patients with adenocarcinoma of unknown primary are excluded
   2. Patients with a diagnosis of two co-existing primary cancers are excluded
10. Abnormal ECGs that are clinically significant such as QT prolongation (QTc > 480 msec), clinically significant cardiac enlargement or hypertrophy, new bundle branch block or existing left bundle branch block, or signs of new, active ischemia a. Patients with evidence of prior infarction who are New York Heart Association (NYHA) functional class II, III, or IV are excluded, as are patients with marked arrhythmia such as Wolff Parkinson White pattern or complete atrioventricular (AV) dissociation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2015-04; Primary Completion 2019-12 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Determination of the safety and tolerability of BBI608 and BBI503 when administered in combination by assessing dose-limiting toxicities (DLTs) | 4 weeks
Determination of the Recommended Phase 2 Dose of BBI608 and BBI503 when administered in combination based on DLT criteria, pharmacokinetic/pharmacodynamic observations and tolerability overall | 20 weeks
  The overall tolerability assessment will include review of persistent grade 2 adverse events and review of adverse events occurring beyond the first cycle.

SECONDARY OUTCOMES:
Pharmacokinetic profile of BBI608 and BBI503 when administered in combination as assessed by maximum plasma concentration and area under the curve. | -5min, 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 hours on day 1, cycles 1 and 2
Pharmacodynamic activity assessed by tumor biopsy | 4 weeks
  Tumor Biopsy to provide information on analysis of the effect of BBI608 and BBI503 on cancer stem cells through immunohistochemistry.
Assessment of the preliminary anti-tumor activity by performing tumor assessments | 16 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Weill Cornell Medical College, New York, New York
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Fort Worth 12th Ave, Fort Worth, Texas
  - Texas Oncology, P.A., San Antonio, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Northwest Cancer Specialists, PC, Vancouver, Washington